CLINICAL TRIAL: NCT01137214
Title: Outcome and Treatment of Complex Sleep Apnea
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Dr. Stephen Corne, University of Manitoba Department of Internal Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2010:026
Record Dates: First submitted 2010-06-01; First posted 2010-06-04 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2010-10

CONDITIONS: Sleep Apnea
Keywords: complex sleep apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CPAP (Active Comparator): Continuous Positive Airway Pressure
  Interventions: Device: Non-invasive positive pressure ventilator
- Adaptive Servo-Ventilator (Active Comparator): Non-invasive positive pressure ventilator that applies a constant expiratory pressure, as well as a variable inspiratory pressure.
  Interventions: Device: Non-invasive positive pressure ventilator

INTERVENTIONS:
Device: Non-invasive positive pressure ventilator — All patients will initially be treated with CPAP for 12 weeks as part of usual clinical treatment for sleep apnea. A sleep study will be conducted after this and prior to randomization into the study. If this repeat sleep study demonstrates persistent central sleep apnea, patients will be randomized into 2 study groups. Group 1 - CPAP for 24 weeks. Group 2 - first 12 weeks CPAP (Continuous Positive Airway Pressure. Next 12 weeks - (ASV) Adaptive Servo ventilation. If the treatment is not working well at 12 weeks the participant/patients have the option of switching to the alternate treatment. Patients will be notified if they are to be switched to ASV. Participants will be asked to fill in the Epworth Sleepiness Score Questionnaire and Sleep Apnea Quality of Life Index form at 12 and 24 weeks.

SUMMARY:
The purpose of the project is:

1. to determine the incidence of complex sleep apnea
2. to determine what percentage of cases will resolve over time with therapy with Continuous Positive Airway Pressure
3. Determine whether there is any difference in outcome, in those with persistent complex sleep apnea on CPAP, between those treated with CPAP or adaptive servo-ventilation.

DETAILED DESCRIPTION:
Patients with suspected obstructive sleep apnea (OSA) are studied overnight in a sleep laboratory, as part of their routine clinical management. If they are found to have OSA during the first half of the night, they are started on continuous positive airway pressure (CPAP) by nasal mask as part of their routine clinical management. A certain percentage of these patients (best estimate from the literature 15%) will develop central sleep apnea (CSA) during their treatment with CPAP.

Participants will be recruited from patients treated with Continuous Positive Airway Pressure (CPAP) for obstructive sleep apnea who develop central sleep apnea (CSA) on CPAP, and are willing to give informed consent .

Patients will be treated with the "best CPAP" pressure, as determined by the sleep physician reading their sleep study. This is defined as the minimum pressure associated with elimination of obstructive events. Patients will be treated with CPAP for 12 weeks. Following treatment, patients will be brought back for a second sleep study to be assessed on CPAP.

Those that demonstrate resolution of CSA on the sleep study will continue on CPAP for an additional 12 weeks. Those that demonstrate persistent CSA will be randomized to either "best CPAP" or Adaptive Servo-ventilation (ASV) therapy for an additional 12 weeks. ASV will be titrated during the second sleep study to determine optimal settings. Patients will be compared at the end of 12 and 24 weeks of treatment regarding response to therapy. This will be assessed by compliance with therapy (as monitored by a smart card within the positive pressure machine), improvement in sleepiness as measured by the Epworth Sleepiness Score, and change in quality of life as measured by the Sleep Apnea Quality of Life Index (SAQLI) a validated quality of life instrument specific to sleep apnea.

In addition, in those who demonstrated persistent central apneas after 12 weeks of CPAP therapy, and were randomized to CPAP or ASV, a third and final sleep study will be done to assess the residual apnea-hypopnea index (the number of respiratory events divided by the number of hours of sleep) on therapy. In those randomized to CPAP who have a persistent poor clinical response associated with an abnormal residual AHI after 24 weeks of treatment, a further 12 week trial of ASV will be undertaken to assess whether it offers any benefit.

In addition to assessing the effect of treatment, the original diagnostic polysomnogram of all patients with complex sleep apnea will be analyzed to determine if there are any polysomnographic features that could be utilized to predict complex sleep apnea before CPAP is applied, (for example: 1) evidence of mixed apneas; or 2) a component of central apneas in addition to the predominant pattern of OSA.)

ELIGIBILITY:
Inclusion Criteria:

* Patient with obstructive sleep apnea who develop central sleep apnea once treated with CPAP

Exclusion Criteria:

* Inability to give informed consent, inability to tolerate positive pressure ventilation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Resolution of sleep apnea | 24 weeks
  As measured by the apnea-hyponea index

SECONDARY OUTCOMES:
Quality of life | 24 weeks
  As measured by Epworth Sleepiness Scale and Sleep Apnea Quality of Life Index

CONTACTS AND LOCATIONS:
Locations (1):
- Miseracordia Sleep Disorders Centre, Winnipeg, Manitoba, Canada